CLINICAL TRIAL: NCT05419479
Title: Phase Ib Open-Label, Multicenter, Study Evaluating the Safety and Efficacy of 'Switch Maintenance' Combination Immunotherapy Using AB154, AB122, and Sotigalimab in Patients With Metastatic Pancreatic Cancer
Brief Title: Switch Maintenance in Pancreatic
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Efficacy concerns.
Sponsor: James Cleary, MD, PhD (Other)
Collaborators: Arcus Biosciences, Inc. (Industry); Lustgarten Foundation (Other)
Responsible Party: Sponsor-Investigator, James Cleary, MD, PhD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-141
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Adenocarcinoma of the Pancreas; Squamous Cell Carcinoma of Pancreas; Adenosquamous Carcinoma of the Pancreas
Keywords: Pancreatic Cancer; Adenocarcinoma of the Pancreas; Squamous Cell Carcinoma of Pancreas; Adenosquamous Carcinoma of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — zimberelimab; sotigalimab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LEAD-IN: DOSE DE-ESCALATION (Experimental): The lead-in dose de-escalation cohort (Phase 1b) will enroll 6 patients (up to 12 patients in 2 dose levels if needed; 6 patients per DL) to receive zimberelimab, domvanalimab, and APX005M
  Interventions: Drug: ZIMBERELIMAB; Drug: DOMVANALIMAB; Drug: APX005M
- ARM A: ZIMBERELIMAB + DOMVANALIMAB + APX005M (Experimental): Participants will be randomly assigned to one of two groups
  Arm A will receive domvanalimab, zimberelimab, and APX005M every two weeks through an infusion.
  Interventions: Drug: ZIMBERELIMAB; Drug: DOMVANALIMAB; Drug: APX005M
- ARM B: FOLFIRI (Active Comparator): Arm B will receive leucovorin, fluorouracil, and irinotecan every two weeks through an infusion
  Interventions: Drug: FOLFIRI
- CROSSOVER: ZIMBERELIMAB + DOMVANALIMAB + APX005M (Experimental): Participants in Arm B (control arm) who experience disease progression (as defined by RECIST v1.1) will be given the option to crossover and receive domvanalimab + zimberelimab, + APX005M in the second-line setting, provided they meet eligibility criteria
  Interventions: Drug: ZIMBERELIMAB; Drug: DOMVANALIMAB; Drug: APX005M

INTERVENTIONS:
Drug: ZIMBERELIMAB — Via IV on two days per cycle, dosage per protocol
  Other Names: AB 122
  Arms: ARM A: ZIMBERELIMAB + DOMVANALIMAB + APX005M; CROSSOVER: ZIMBERELIMAB + DOMVANALIMAB + APX005M; LEAD-IN: DOSE DE-ESCALATION
Drug: DOMVANALIMAB — Via IV on two days per cycle, dosage per protocol
  Other Names: AB 154
  Arms: ARM A: ZIMBERELIMAB + DOMVANALIMAB + APX005M; CROSSOVER: ZIMBERELIMAB + DOMVANALIMAB + APX005M; LEAD-IN: DOSE DE-ESCALATION
Drug: APX005M — Via IV on two days per cycle, dosage per protocol
  Other Names: CD40
  Arms: ARM A: ZIMBERELIMAB + DOMVANALIMAB + APX005M; CROSSOVER: ZIMBERELIMAB + DOMVANALIMAB + APX005M; LEAD-IN: DOSE DE-ESCALATION
Drug: FOLFIRI — every two weeks through an infusion at a dose determined by physician
  Arms: ARM B: FOLFIRI

SUMMARY:
This study is being done to test the safety and effectiveness of combining domvanalimab (AB154), zimberelimab (AB122), and APX005M with pancreatic cancer that has spread to other parts of body.

This research study involves immunotherapy. Immunotherapy triggers the body's immune system to fight cancer cells.

The names of the study drugs involved in this study are:

* Domvanalimab (also known as AB154)
* Zimberelimab (also known as AB122)
* APX005M

DETAILED DESCRIPTION:
This is an open-label, Phase 1b/2, multicenter, randomized study evaluating the safety and efficacy of 'switch maintenance' combination immunotherapy (domvanalimab) zimberelimab and APX005M versus 'continuous maintenance' in patients with metastatic pancreatic cancer following 4-6 months of FOLFIRINOX

The names of the study drugs involved in this study are:

* Domvanalimab (also known as AB154)
* Zimberelimab (also known as AB122)
* APX005M

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will be randomized into one of two groups:

* Arm A will receive domvanalimab, zimberelimab, and APX005M every two weeks through an infusion.
* Arm B will receive leucovorin, fluorouracil, and irinotecan every two weeks through an infusion

If you are in Arm B and the drugs stop working, participants may receive the drugs given in Arm A.

Participants will receive study treatment as long the disease does not worsen or there are no serious side effects for a maximum of 26 cycles (2 years) and will be followed for 12 months after the discontinue the study drugs.

It is expected that about 46 people will take part in this research study.

This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational drug or drugs and also tries to define the appropriate dose of the investigational drug(s) to use for further studies. Phase II clinical trials test the safety and effectiveness of an investigational drug or drugs to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved domvanalimab, zimberelimab, or APX005M as a treatment for any disease.

drug regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed pancreatic cancer (adenocarcinoma, squamous, or adenosquamous histologies) that is metastatic and for which standard curative or palliative measures do not exist or are no longer effective. Locally advanced patients are not eligible.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
* Participants must have received 8-12 cycles (4-6 months) of first-line FOLFIRINOX or modified FOLFIRINOX with stable disease or better.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of domvanalimab + zimberelimab + APX005M in participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤1
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), except in patients with documented Gilbert's syndrome, who must have a total bilirubin ≤ 3 x ULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x institution's upper limit of normal (ULN) for patients with no concurrent liver metastases, OR ≤ 5.0 x institution's ULN for patients with concurrent liver metastases creatinine OR glomerular filtration rate (GFR) creatinine ≤ 2 x ULN OR GFR measured by calculated creatinine clearance (CrCl) > 45 mL/min. CrCl can be calculated using the Cockroft-Gault method.
  * Hemoglobin (Hgb) >9.0 g/dL
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. If a participant has brain or meningeal metastases, the participant must meet the following criteria:

  * Have no evidence of progression by neurologic symptoms or sign for at least 4 weeks prior to the first dose.
  * Metastatic brain lesions do not require immediate intervention.
  * Carcinomatous meningitis is excluded regardless of clinical stability.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Participants must be willing to undergo a pre-treatment fresh tumor biopsy.
* Participants must be willing to undergo an on-treatment tumor biopsy (if medically feasible).
* Participants must have archival tissue available for analysis, which will be used for correlative studies if a pretreatment biopsy reveals necrotic tissue.

  * The effects of domvanalimab, zimberelimab, and APX005M on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (See Section 5.6) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of domvanalimab, zimberelimab, or APX005M administration.
  * Women of childbearing potential (WOCBP), defined as not surgically sterilized and between menarche and 1-year post menopause, must have a negative serum pregnancy test within 7 days prior to the first dose of investigational therapies and a negative urine (or serum) pregnancy test within 3 days prior to the first dose of investigational therapies.
  * WOCBP must agree to use highly effective methods of contraception from the time of consent, through the duration of study treatment, and 5 months after the last dose of investigational therapies.
  * Male participants with WOCBP sexual partners must agree to use highly effective methods of contraception, and to refrain from donating sperm from the time of consent through the duration of study treatment and 7 months after the last dose of investigational therapies. Contraceptive requirements may be extended depending on local regulatory requirements.
  * Female participants must not be breast feeding and must not breast-feed a baby while on treatment and for up to 7 months after the last dose of investigational therapies.
* Ability to understand and the willingness to sign a written informed consent document.
* Willing and able to comply with the requirements and restrictions in this protocol.
* Eligibility Criteria for Stage 2 (Crossover Stage)

  * Patients must meet all of the criteria used for Stage 1.
  * Patients allocated to the control arm (Arm B) during Stage 1 have the ability to initiate Stage 2 treatment within 4 weeks after experiencing disease progression per RECIST v1.1 while receiving control treatment
* Availability of a tumor specimen from on-treatment biopsy during Expansion Phase. If this is not available, willingness to undergo biopsy prior to initiation of Crossover Phase.
* Exclusion Criteria (for both Stage 1 and Stage 2)
* Patients who have evidence of disease progression on FOLFIRINOX.
* Participants who have had cytotoxic chemotherapy, radiotherapy, within 2 weeks prior to the first dose of study medication or those who have not recovered to ≤ CTCAE Grade 1 or baseline from adverse events due to agents administered more than 2 weeks earlier. Exceptions include alopecia of any grade and Grade ≤ 2 peripheral neuropathy.
* Participants who have received any other investigational agents for pancreatic cancer.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies, or allergic reactions attributed to compounds of similar chemical or biologic composition to domvanalimab, zimberelimab, APX005M, or other agents used in study.
* Prior treatment with any of the protocol-specified study treatments, with the exception of chemotherapy.
* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies (including anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-TIGIT, and CD40 agonist therapeutic antibodies)
* Patients with endocrine or acinar pancreatic carcinoma are not eligible for the study.
* Known dihydropyrimidine dehydrogenase deficiency.
* Patients who are enrolling after achieving at least stable disease on FOLFIRINOX are not eligible if they have a germline BRCA1 or BRCA2 mutation(s).
* Participants who have undergone major surgery 28 days prior to initiating protocol therapy. Participants must have sufficiently recovered from adverse events caused by the procedure as judged by the treating investigator. Placement of central venous access catheter (e.g., port or similar) is not considered a major surgical procedure.
* Participants must not have a history of human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV), except for the following:

  * Participants with anti-HepB core antibody but with undetectable HepB virus deoxyribonucleic acid (DNA) and negative for HepB surface antigen
  * Participants with resolved or treated hepatitis C virus (HCV) (i.e., HCV antibody positive but undetectable HCV RNA)
* Participants must not have a history of primary immunodeficiency.
* Active autoimmune disease, history of autoimmune disease, or concurrent administration of immune suppressive medications. Participants must not have a known or suspected history of an autoimmune disorder within 3 years of the first dose of investigational agent, including but not limited to: systemic lupus erythematosus, scleroderma, inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, sarcoidosis, or autoimmune hepatitis. Exceptions include participants with Type 1 diabetes mellitus, hypothyroidism requiring only hormone replacement, skin disorders such as alopecia or vitiligo, not requiring systemic therapy, resolved childhood asthma/atopy, or conditions not expected to recur in the absence of an external trigger are eligible. Patients with a history of Hashimoto syndrome within 3 years of the first dose of investigational agent, which resolved to hypothyroidism alone.
* Prior allogeneic bone marrow transplantation or solid organ transplantation.
* Participants must not receive concurrent or prior use of an immunosuppressive agent within 14 days prior to the first dose of investigational agent. Exceptions include:

  * Systemic steroids at physiologic doses (equivalent to dose of ≤ 10 mg oral prednisone) are permitted.
  * Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
  * Patients with a condition with anticipated use of systemic steroids above the equivalent of 10 mg prednisone are excluded.
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Patients must not have received a live attenuated vaccine within 28 days before the first dose of investigational agent, and patients, if enrolled, should not receive live vaccines during the study or for 180 days after the last dose of investigational agent. Prior COVID-19 infection and/or COVID-19 vaccination is permitted.
* Known hereditary or acquired coagulopathy (e.g., hemophilia, von Willebrand disease, cancer-associated diffuse intravascular coagulation)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (viral, bacterial, or fungal infections requiring parenteral treatment within 14 days of the initiation of investigational therapy), clinically significant cardiovascular disease, unstable angina pectoris, cardiac arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with a history of a clinically relevant second primary malignancy within the past 2 years. Exceptions include: resected basal and squamous cell carcinomas of the skin and completely resected carcinoma in situ of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities-Phase 1 | 28 Days
  Toxicity assessments will be evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Every 8 weeks up to 38 Months
  Tumor reassessment with baseline CT scan and restaging scans will occur every 8 weeks using RECIST v1.1
Disease Control Rate | Every 8 weeks up to 38 Months
  Tumor reassessment with baseline CT scan and restaging scans will occur every 8 weeks using RECIST v1.1
Switch Maintenance-Progression Free Survival | baseline up to 38 months
  PFS will also be measured for post-Folfirinox (PFS2). PFS is defined as the time from registration to the Crossover Arm to the earlier of progression or death due to any cause.
  The PFS2 distribution will be calculated and plotted using the Kaplan-Meier method
Duration of Response (DoR) | Baseline up to 38 Months
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Overall Survival | baseline up to 38 months
  Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive
Number of Participants With Treatment-Related Adverse Events | Up to 38 Months
  Toxicity assessments will be evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: James Cleary, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu